CLINICAL TRIAL: NCT03529370
Title: Sonography of the Optic Nerve Sheath Diameter for Detection of Elevated Intracranial Pressure Compared to Computed Tomography
Brief Title: Sonography of the Optic Nerve Sheath Diameter for Detection of Elevated Intracranial Pressure (ICP)
Status: Completed | Type: Observational
Sponsor: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Islam Hassan Mohamed Elsadek Abulnaga, Specialist of critical care medicine, National heart institute, Cairo, Egypt, National Heart Institute, Egypt
Other Study IDs: Optic nerve sonography and ICP
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Intracranial Hypertension
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: optic nerve ultrasound — sonograhy of the optic nerve sheath diameter

SUMMARY:
In this study the invistigators chose to measure the optic nerve sheath diameter by sonography for diagnosis of elevated intracranial pressure (ICP) in comparison to brain computed tomograhy (CT) as the reference gold standard for detection of raised ICP since optic nerve songraphy is radiation-free , noninvasive, and has certain features which increase its convenience portability, easy application, low cost, repeatability on request, bedside application, short application time and applicability even in the presence of unstable vital signs.

DETAILED DESCRIPTION:
Elevated intracranial pressure (ICP) is seen in head trauma, hydrocephalus, intracranial tumors, hepatic encephalopathy, and cerebral edema. Intractable elevated ICP can lead to death or devastating neurological damage either by reducing cerebral perfusion pressure (CPP) and causing cerebral ischemia or by compressing and causing herniation of the brainstem or other vital structures. Prompt recognition is crucial in order to intervene appropriately.

Intractable high ICP is the most common "terminal event" leading to death in neurosurgical patients. The association between the severity of intracranial hypertension and poor outcome after severe head injury is well recognized. Outcomes tend to be good in patients with normal ICP, whereas those with elevated ICP are much more likely to have an unfavorable outcome. Elevated ICP carries a mortality rate of around 20%.

The rapid recognition of elevated ICP is therefore of obvious and paramount importance so that it can be monitored and so that therapies directed at lowering ICP can be initiated. A raised ICP is measurable both clinically and quantitatively. Continuous ICP monitoring is important both for assessing the efficacy of therapeutic measures and for evaluating the evolution of brain injury.

The goal of ICP monitoring is to ensure maintenance of optimal CPP. The ICP also forms a basis for medical or surgical intervention in cases of increased ICP with agents such as 3% sodium chloride (NaCl), mannitol, or diuretics (Loop diuretics), ventriculostomy, cerebrospinal fluid (CSF) diversion, and phentobarbital coma or surgical decompression in cases of intractable ICP elevation that do not respond to conservative management.

ICP monitoring may be discontinued when the ICP remains in the normal range within 48-72 hours of withdrawal of ICP therapy or if the patient's neurological condition improves to the point where he or she is following commands.

Since many investigators have questioned invasive ICP monitoring in improving patient outcomes, the invistigators tried to find noninvasive method of ICP monitoring.

The optic nerve sheath is contiguous with the dura mater, and its contents are contiguous with the subarachnoid space. Thus, raised intracranial pressure (ICP) leads to an increase in the optic nerve sheath diameter.

A-mode sonography was first used for visualization of the optic nerve sheath; however, it was not until 1994, when Hansen et al used B-mode sonography, when the approach to measurement was standardized. Sonographic studies of cadaveric optic nerves together with the work of Hansen et al established that the greatest degree of distension of the sheath occurred 3 mm behind the optic globe. This location has become the standard measurement point.

As a technique, ocular sonography is quickly learned; Tayal et al showed that with an experienced operator, 10 scans with 3 abnormal scans should be sufficient training, whereas in new ultrasound operators, 25 may be needed. In addition to these findings, measurement of both eyes can be performed in less than 4 minutes.

the invistigators chose CT as the reference gold standard for detection of raised ICP as simple noninvasive method in critically ill patients. Raised ICP is diagnosed with CT on a daily basis in clinical practice. Treatments are initiated, hemicraniectomies are performed, and intraventricular shunts are inserted, all on the basis of raised ICP as seen on imaging.

The findings of elevated ICP in cranial CT (CCT) include:

1. changes in ventricular sizes;
2. lessening in basilar cistern sizes;
3. narrowing or eliminating in sulci;
4. transfalcine herniation; and
5. changes in the rate of grey/white matter. So in this study the invistigators chose to measure optic nerve sheath diameter by sonography for diagnosis of elevated ICP in comparison to brain CT as the reference gold standard for detection of raised ICP

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected raised ICP such as:

  1. Patients with traumatic brain injury
  2. Patients with intracranial tumours
  3. Patients with hepatic encephalopathy
  4. Cerebral edema: Due to head injury, ischemic stroke with vasogenic edema, hypoxic or ischemic encephalopathy, postoperative edema

Exclusion Criteria:

* Patients with edema or trauma in the eye lid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult patients with clinically suspected raised ICP such as:
  1. Patients with traumatic brain injury
  2. Patients with intracranial tumours
  3. Patients with hepatic encephalopathy
  4. Cerebral edema: Due to head injury, ischemic stroke with vasogenic edema, hypoxic or ischemic encephalopathy, postoperative edema
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
To measure the optic nerve sheath diameter by optic nerve ultrasound in patients with elevated ICP before and after osmotherapy and to measure the accuracy of occular ultrasound in diagnosis of elevated ICP compared to cranial computed tomography (CT) | up to 48 hours
  Cranial CT and optic nerve US will be done once elevated ICP is suspected clinically to find signs of elevated ICP in cranial CT and measure the optic nerve sheath diameter by optic nerve ultrasound and then follow up optic nerve sonograhy and cranial CT will be done after 48 hours of giving osmotheray to detect the effect of osmotherapy on signs of elevated ICP in cranial CT and on the optic nerve sheath diameter

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Abdallah, MD, Study Director — Cairo University; Suzy F Michael, MD, Study Director — Cairo University; Hassan K Nagi, MD, Study Director — Cairo University
Locations (1):
- National heart institute , Imbaba, Cairo, Egypt

REFERENCES:
- [Background] Robba C, Cardim D, Tajsic T, Pietersen J, Bulman M, Rasulo F, Bertuetti R, Donnelly J, Xiuyun L, Czosnyka Z, Cabeleira M, Smielewski P, Matta B, Bertuccio A, Czosnyka M. Non-invasive Intracranial Pressure Assessment in Brain Injured Patients Using Ultrasound-Based Methods. Acta Neurochir Suppl. 2018;126:69-73. doi: 10.1007/978-3-319-65798-1_15. PMID 29492535
- [Background] Wang LJ, Chen LM, Chen Y, Bao LY, Zheng NN, Wang YZ, Xing YQ. Ultrasonography Assessments of Optic Nerve Sheath Diameter as a Noninvasive and Dynamic Method of Detecting Changes in Intracranial Pressure. JAMA Ophthalmol. 2018 Mar 1;136(3):250-256. doi: 10.1001/jamaophthalmol.2017.6560. PMID 29392301